CLINICAL TRIAL: NCT04497246
Title: Psychological Impact, Mental Health and Sleep Disorder Among Patients Hospitalized and Health Care Workers During the 2019 Coronavirus Outbreak (COVID-19)
Status: Completed | Type: Observational
Sponsor: Murielle Surquin (Other)
Responsible Party: Sponsor-Investigator, Murielle Surquin, Head of geriatry department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHU-COVIDIMPACT
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly patients: Elderly patients (over 65 years old) hospitalized for COVID-19 within the CHU Brugmann Hospital
  Interventions: Other: Questionnaire
- Health Care professionals: Health Care professionals working within the CHU Brugmann Hospital
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Data collection by means of various questionnaires

SUMMARY:
COVID-19 is an infectious disease caused by the last coronavirus discovered, called SARS-CoV-2. Symptoms encountered in COVID-19 are: cough, breathing difficulties (dyspnea, chest pain, etc.), pyrexia, anosmia (loss of smell) and/or dysgeusia (loss of taste), but also ENT symptoms (rhinitis type, odynophagia), headaches, asthenia, muscle pain, confusion and diarrhea. Infection with SARS-CoV-2 can also be asymptomatic. COVID-19 can be passed from person to person by respiratory droplets expelled when a person speaks, coughs or sneezes. The currently estimated incubation period ranges from 1 to 14 days, and most often this is around 5 days.

According to a literature review, there is strong evidence that COVID-19 has an impact on mental health (anxiety being the most common symptom) whether in the general population, healthcare workers or vulnerable populations. The objective of this project is to assess mental health and sleep disorders within two populations: elderly patients and nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 65 years of age or older, having been hospitalized for COVID-19 within the CHU Brugmann Hospital
* People aged 18 or over, member of the nursing staff of the CHU Brugmann Hospital, having worked during COVID-19.

Exclusion Criteria:

* Incoherent patients
* Severe presbycusis
* Oral expression impairment
* Insurmountable language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Subjects 65 years of age or older, having been hospitalized for COVID-19 within the CHU Brugmann Hospital
  * People aged 18 or over, member of the nursing staff of the CHU Brugmann Hospital, having worked during COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Impact Event Scale-Revised (IES-R) | 15 minutes
  The IES-R is a 22-item self-report measure that assesses subjective distress caused by traumatic events.Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales.
Generalised Anxiety Disorder-7 (GAD-7) | 15 minutes
  Self-administered patient questionnaire used as a screening tool and severity measure for generalised anxiety disorder (GAD).The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Patient Health Questionnaire-9 (PHQ-9) | 15 minutes
  The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care. It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment.
Insomnia severity index (ISI) | 15 minutes
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia.The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

SECONDARY OUTCOMES:
Demographic data | 1 year
  Age, gender, familial status, home status (living alone/family support/healthcare support/ retirement home).
Hospitalization duration | 1 year
  Hospitalization duration
ICU stay | 1 year
  Hospitalization within the intensive care unit (yes/no) with or without intubation
Medical history | 1 year
  History of chronic diseases
Alcohol consumption | 1 year
  Alcohol consumption : none - stable - increased - diminished
Tobacco consumption | 1 year
  Tobacco consumption : none - stable - increased - diminished

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Levy, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No